CLINICAL TRIAL: NCT03873766
Title: Management of Pleural Space Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY2018000278
Record Dates: First submitted 2018-10-02; First posted 2019-03-13 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Empyema, Pleural; Parapneumonic Effusion
MeSH Terms: conditions — Empyema, Pleural | interventions — Surgical Procedures, Operative; Quality of Life

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either IPFT or surgery for treatment of their complex pleural space infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intrapleural fibrinolytic therapy (IPFT) (Active Comparator): * Procedure/Surgery: Pleural Sampling
  * Procedure/Surgery: Pleural fluid drainage
  * Protocol Image #1: After chest tube is placed, imaging is obtained within 24-48 hours to assess the fluid drainage.
  * Other: Surgical Consultation
  * Intrapleural Medications (IPFT): The IPFT group will receive a total of 5-6 doses of alteplase 10mg and DNase 5 mg twice daily x 3 days. delivered through a chest tube or small bore catheter into the pleural space. The doses will be given twice a day.
  * Protocol Image #2: Chest X-ray PA/Lateral: The morning after intervention completion, a chest X-ray PA/lateral will be obtained
  * Quality of Life: Quality of life will be measured at 30 day and 90 day and 1 year clinical follow-up using the SF-36 quality of life survey and return to work questionnaires
  Interventions: Drug: Intrapleural Medications; Procedure: Pleural Sampling; Procedure: Pleural fluid drainage; Radiation: Protocol Image #1; Other: Surgical Consultation; Radiation: Protocol Image #2: Chest X-ray PA/Lateral; Behavioral: Quality of Life
- Surgery (Active Comparator): * Procedure/Surgery: Pleural Sampling
  * Procedure/Surgery: Pleural fluid drainage: Chest tube placement
  * Protocol Image #1: Once the chest tube is placed, imaging is obtained within 24-48 hours to assess the fluid drainage.
  * Other: Surgical Consultation
  * Surgery: The surgical arm will have either open surgery or a VATS approach at the discretion of the surgeon
  * Protocol Image #2: Chest X-ray PA/Lateral: The morning after intervention completion (surgery or last dose of IPFT), a chest X-ray PA/lateral will be obtained
  * Quality of Life: Quality of life will be measured at 30 day and 90 day and 1 year clinical follow-up using the SF-36 quality of life survey and return to work questionnaires
  Interventions: Procedure: Surgery; Procedure: Pleural Sampling; Procedure: Pleural fluid drainage; Radiation: Protocol Image #1; Other: Surgical Consultation; Radiation: Protocol Image #2: Chest X-ray PA/Lateral; Behavioral: Quality of Life

INTERVENTIONS:
Drug: Intrapleural Medications — The IPFT group will receive a total of 5-6 doses of alteplase 10mg and DNase 5 mg twice daily x 3 days. delivered through a chest tube or small bore catheter into the pleural space. The doses will be given twice a day. If the first IPFT dose is given in the evening on the first day, they will only receive a total of 5 doses of the dual-agent IPFT (alteplase and DNase).
  Other Names: IPFT
  Arms: Intrapleural fibrinolytic therapy (IPFT)
Procedure: Surgery — The surgical arm will have either open surgery or a Video assisted Thoracoscopic Surgery (VATS) approach at the discretion of the surgeon
  Arms: Surgery
Procedure: Pleural Sampling — Pleural fluid may be sampled by the responsible clinical service in the course of clinical care for patients with suspected pulmonary infection or by consulting service after identification of patient. Some patients will have a thoracentesis or tube drainage, and others will have no intervention at the time of referral for study eligibility review. Enrollment reflects real world clinical care and patients will be considered for enrollment regardless of sampling techniques or timing prior to evaluation
Procedure: Pleural fluid drainage — All patients in the study must have tube thoracostomy for drainage of the pleural space. This may have been done by the clinically responsible team or by the study team. Physicians may select chest tubes of any type, but the minimum size is 14 French. For patency, chest tubes 14-20 French should be kept at negative 20 suction and flushed daily. Large bore chest tubes (>20French) may be kept at negative 20 suction at the discretion of the physician managing the chest tube and do not require daily flushing. Supportive care will follow Institutional Guidelines.
Radiation: Protocol Image #1 — Once the chest tube is placed, imaging is obtained within 24-48 hours to assess the fluid drainage. The choice of image, either Chest X-ray or CT Chest, is up to the discretion of the treating physician. Based on the imaging, patients will be separated into 2 groups:
  A: Complete drainage/re-expansion of the lung: If there is complete drainage of the pleural fluid collection and lung re-expansion based on image #1, patients will follow usual clinical care without randomization and be observed until discharge. Patients will remain in the study and their data will be collected.
  B: Incomplete drainage/incomplete lung re-expansion: For those patients that have incomplete drainage of the pleural fluid collection on image #1 and/or the lung does not re-expand.
Other: Surgical Consultation — A thoracic surgery consultation will be obtained on all patients with incomplete drainage and/or the lung does not re-expand, to determine surgical candidacy. Those patients that the surgical team deem unsafe for surgery will receive clinically appropriate guideline centered, non-surgical, care. These patients will not be randomized but they will remain in the study and their data will be collected. Criteria deeming patients unfit for surgery include, but are not limited to: inability to tolerate single lung ventilation, severe chronic obstructive pulmonary disease (COPD), and risk of surgery prohibitive. Patients not excluded from surgery will be randomized.
Radiation: Protocol Image #2: Chest X-ray PA/Lateral — The morning after intervention completion (surgery or last dose of IPFT), a chest X-ray PA/lateral will be obtained (protocol image #2). Based on Image #2 the patient will be categorized into one of three groups: satisfactory improvement of pleural fluid collection, unsatisfactory improvement in pleural fluid collection on imaging, or treatment failures.
Behavioral: Quality of Life — Quality of life will be measured at 30 day and 90 day and 1 year clinical follow-up using the SF-36 quality of life survey and return to work questionnaires

SUMMARY:
Currently, there is no high-quality evidence comparing the clinical outcomes and cost effectiveness of surgical drainage combined with antibiotics versus dual-agent intrapleural fibrinolytic therapy (IPFT) catheter drainage of pleural space infections with concomitant antibiotic therapy. The absence of comparative data is a challenge for surgical and medical services in clinical decision-making for this common and morbid condition.

This is a pilot study comparing surgical drainage of the pleural space in complex pleural effusions to bedside chest tube drainage using dual agent IPFT with the intent to inform on study algorithm and endpoint performance in anticipation of a multi-institutional randomized clinical trial.

DETAILED DESCRIPTION:
Currently, there is no high-quality evidence comparing the clinical outcomes and cost effectiveness of surgical drainage combined with antibiotics versus dual-agent intrapleural fibrinolytic therapy (IPFT) catheter drainage of pleural space infections with concomitant antibiotic therapy. The absence of comparative data is a challenge for surgical and medical services in clinical decision-making for this common and morbid condition.

This is a pilot study comparing surgical drainage of the pleural space in complex pleural effusions to bedside chest tube drainage using dual agent IPFT with the intent to inform on study algorithm and endpoint performance in anticipation of a multi-institutional randomized clinical trial.

Patient's with complex pleural space infections identified at the institution that meet inclusion criteria will be randomized to receive either IPFT or surgical debridement after a surgery consultation is obtained. Patients randomized to the IPFT study arm will receive a total of 5-6 doses of alteplase 10mg and DNase 5 mg BID x 3 days delivered through a chest tube or small bore catheter into the pleural space. The doses will be given twice a day. If the first IPFT dose is given in the evening on the first day, they will only receive a total of 5 doses of the dual-agent IPFT (alteplase and DNase). The surgical arm will have either open surgery of a VATS approach at the discretion of the surgeon.

IPFT (alteplase and DNase) is not an investigational agent. It is used in standard of care practice for the treatment of complex pleural space infections. The investigators seek to compare dual-agent IPFT (alteplase and DNase) to surgery in this study. As such, the IPFT agents will be ordered from pharmacy through the electronic medical record (EMR) as in normal practice and there is not a study drug.

After drainage, patients will be followed with protocol images to assess the drainage of their pleural space. If there is satisfactory improvement in the pleural fluid collection on imaging chest tube or small bore catheter will be removed per protocol in both study arms. Chest tube removal protocol is based on fluid character and measured output.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinical presentation compatible with pleural infection (fever or leukocytosis, elevated procalcitonin, elevated C-reactive protein (CRP))
* Pleural fluid requiring drainage that is either:

  * Macroscopically purulent or
  * Positive on culture for bacterial infection or
  * Positive for bacteria on gram stain or
  * Lactate dehydrogenase (LDH) > 1000 IU/L or
  * Glucose <40 mg/dL

Exclusion Criteria:

* Age <18 years
* Unable to give consent (No surrogate consent of legally authorized representatives allowed for this study)
* Not proficient in English
* History of prior ipsilateral empyema
* Has known sensitivity to DNase or alteplase
* History of intracranial hemorrhage or acute intracranial hemorrhage
* History of stroke, hemorrhage, or trauma within the last 3 months
* Has had prior surgery on the side of the pleural infection
* Patients who are pregnant or lactating
* Expected survival less than 6 months from a different pathology to this pleural infection based on clinical judgment
* Has a tunneled pleural catheter in place
* Patients on anticoagulation that cannot be interrupted for surgical intervention
* Patients with known or suspected malignant pleural effusion
* Patients with renal failure (Creatinine clearance <30)
* Prior history of or concern for chylothorax or pseudochylothorax
* Vulnerable populations: prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of the proposed study algorithm as measured by percent of subjects enrolled to study completion, percent of subjects randomized but did not complete the study, and percent of health care professional protocol deviation | From patient identification to 1 year post discharge
  • Test the feasibility of the proposed study algorithm to compare Intrapleural fibrinolytic therapy (IPFT) to surgical intervention as measured by percent enrollment to completion of study algorithm and multidisciplinary participation in adherence to the algorithm.
Subject identification and accrual as measured by the percent of patients not screened and randomized and the time to accrual of 20 patients of the number of patients accrued in one year | From patient identification to 1 year post discharge
  Subject identification and accrual as measured by the percent of patients not screened and randomized and the time to accrual of 20 patients of the number of patients accrued in one year

SECONDARY OUTCOMES:
Radiographic improvement | From date of protocol Image #1 (once the chest tube is placed, protocol image #1 is obtained within 24-48 hours) to date of protocol Image #2 (the morning after intervention, approximately 12-24 hours after intervention)
  Imaging will be posterior-anterior (PA) and lateral chest x-ray to determine radiographic change. Images will be saved and exported as JPEG files and opened in image editing software. Polygons will be drawn representing fluid collections and the hemithorax area covered will be calculated with the volume derived.
  Change in fluid volume will be quantified as:
  * Less than 50%
  * Between 50-75%
  * Greater than 75% Change of greater than 75% will be considered satisfactory improvement. Chest radiograph images will be reviewed and measured by two independent radiologists. If greater than 5% discrepancy in fluid volume change is reported, the independent radiologists will re-read and re-measure the images together.
Number of participants who have treatment failures needing further treatment crossover (IPFT to surgery; surgery to IPFT) | From patient identification to 1 year post discharge
  Treatment failures are defined as any patients with evidence of ongoing infection, persistently undrained pleural space and fever or elevated inflammatory markers still present at least 48 hours after completion of their intervention. Treatment failures will be treated at the discretion of the clinically responsible team, this may include but is not limited to study arm crossover. If a patient is a treatment failure and has treatment crossover (IPFT to surgery, surgery to IPFT), the data will documented with the data collection.
Number of participants with procedure related complications | From intervention with IPFT or surgery to date of discharge from hospital, usually 7-10 days
  Documented using the Common Terminology Criteria for Adverse Events (CTCAE)
Quality of life Surveys: 36-Item Short Form Survey (SF-36) | Quality of life will be measured at 30 day and 90 day clinical follow-up
  Quality of life will be measured at 30 day and 90 day clinical follow-up using the SF-36 quality of life survey. The SF-36 is a 36 question survey that assesses survey general health on a scale of 1-5 (1=excellent, 5=poor). In addition it assesses how current health limits activities such as walking, daily activities of bathing and dressing oneself. A higher score defines a more favorable health state. Each item is score on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Secondarily, the scores to each question are averaged in the groups in which they are categorized to create an 8 scale scores. The 8 scale categories are: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health.
Cost comparison | From date of intervention with IPFT or surgery to date of discharge from hospital, usually 7-10 days
  Cost Comparison: As one of the secondary endpoints for the study, we will perform a cost comparison between the two study arms (IPFT and surgical drainage). Cost data will be obtained from billing data from the patient's hospital admission for stay and procedures related to the patients complicated pleural space infection. No billing data will be obtained directly from the participants in the study.
Chest tube duration | From date of initiation of intervention of IPFT or surgery (approximately 24-48 hours after patient identification) to date of removal of chest tube, approximately 7 days after placement depending on the intervention and the chest tube output.
  The length of time the chest tube is in the patient. The study algorithm governs chest tube removal parameters: Once it has been deemed that there is satisfactory improvement in imaging and no signs of ongoing infection, the chest tube will be removed per protocol. Criteria for removal: Fluid non purulent, serous in character, pleural drain output is less than 200 cc/24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jed Gorden, MD, Principal Investigator — Swedish Cancer Institute
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilshire CL, Jackson AS, Vallieres E, Bograd AJ, Louie BE, Aye RW, Farivar AS, White PT, Gilbert CR, Gorden JA. Effect of Intrapleural Fibrinolytic Therapy vs Surgery for Complicated Pleural Infections: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e237799. doi: 10.1001/jamanetworkopen.2023.7799. PMID 37043201